CLINICAL TRIAL: NCT03030911
Title: The Effect of Dexmedetomidine vs Midazolam on Resting Energy Expenditure in Critically Ill Patients: Randomized Controlled Study
Brief Title: Dexmedetomidine vs Midazolam on Resting Energy Expenditure in Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Lecturer of anesthesia and critical care medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N-26-2016
Record Dates: First submitted 2017-01-19; First posted 2017-01-25 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Mechanical Ventilation; Dexmedetomidine; Midazolam; Sedation
MeSH Terms: interventions — Dexmedetomidine; Midazolam; Fentanyl; Calorimetry, Indirect; Calorimetry

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Active Comparator): * Patients will receive analgesia with fentanyl at a ﬁxed dose of 1 µg.kg.hr-1. Each patient will receive the study drug within 24 hours after intubation. Sedatives used before study enrolment will be discontinued 6 hours prior to the initiation of study drug.
  * Group I patients will have dexmedetomidine (0.075 µg.kg-1.mL-1). Dexmedetomidine infusion will be started at 0.15 µg.kg-1.hr-1 (2 mL.hr-1) and will be adjusted by 0.15 µg.kg-1.h-1 increments to a maximum of 0.75 µg/kg/h (10 ml.h-1)
  * Intervention: indirect calorimetry
  Interventions: Drug: Dexmedetomidine; Drug: Fentanyl; Device: Indirect calorimetry
- midazolam group (Placebo Comparator): * Patients will receive analgesia with fentanyl at a ﬁxed dose of 1 µg.kg.hr-1. Each patient will receive the study drug within 24 hours after intubation. Sedatives used before study enrolment will be discontinued 6 hours prior to the initiation of study drug.
  * Group II patients will have midazolam (0.5 mg.mL-1). Midazolam will be started at 1 mg.h-1 (2 mL.hr-1) and adjusted by 1 mg.h-1 to a maximum of 5 mg.h-1 (10 mL.h-1). All infusions will be adjusted by increments of 2 mL.hr-1 to maintain blinding. Patients in either group not adequately sedated by the maximum infusion rate of the study medication will receive a bolus dose of fentanyl 0.5 µg.kg-1.
  * Intervention: indirect calorimetry
  Interventions: Drug: Midazolam; Drug: Fentanyl; Device: Indirect calorimetry

INTERVENTIONS:
Drug: Dexmedetomidine — The drug will be administered for sedation and its effect on basal metabolic rate will be investigated
  Other Names: Precedex
  Arms: Dexmedetomidine group
Drug: Midazolam — The drug will be administered for sedation and its effect on basal metabolic rate will be investigated
  Other Names: dormicum
  Arms: midazolam group
Drug: Fentanyl — The drug will be administered in both groups
Device: Indirect calorimetry — The device will be used for measurement of basal metabolic rate
  Other Names: Calorimetry

SUMMARY:
The aim of this study is to compare the effect of dexmedetomidine on resting energy expenditure in relation to the midazolam in critically ill patients using indirect calorimetry

DETAILED DESCRIPTION:
Caloric needs in critically-ill patients fluctuate significantly over the course of the disease which might expose patients to either malnutrition or overfeeding. Malnutrition is associated with deterioration of lean body mass, poor wound healing, increased risk of nosocomial infection, and weakened respiratory muscles. On the other hand overfeeding in medically compromised patients can promote lipogenesis, hyperglycemia, and exacerbation of respiratory failure. Many factors may affect the resting energy expenditure (REE) through manipulation of oxygen consumption (VO2).

Sedatives are important contributors to reduction of REE. The postulated mechanism of sedative-induced reduction of VO2 is inhibition of circulating catecholamine and pro-inflammatory cytokines.

Dexmedetomidine is a highly selective α2-adrenoceptor agonist. Stimulation of the α2-adrenoceptor in the central nervous system causes a 60-80% reduction in sympathetic outflow and endogenous catecholamine levels. It was found that perioperative use of α2 agonists decreased sympathetic activity with subsequent reduction of VO2 and REE. Moreover, dexmedetomidine, has some anti-inflammatory effect by inhibiting the pro-inflammatory cytokines which may cause additional reduction of REE in critically ill patient.

Midazolam is another important sedative that is frequently used in critically-ill patient. Terao et al. found that increasing the depth of sedation using midazolam, decreased oxygen consumption and REE. However, it remains unclear whether the effect of midazolam on REE is related to the drug itself or to the depth of sedation.

There is no direct comparison in the literature between dexmedetomidine and midazolam on REE.

ELIGIBILITY:
Inclusion Criteria:

* The study will be designed to recruit 30 critically-ill patients who will be admitted to the surgical ICU for ventilatory support and will be expected to continue for 2 days or longer.

Exclusion Criteria:

* Age < 18 years old.
* Pregnant patient.
* Serious central nervous system pathologies (traumatic brain injury, acute stroke, uncontrolled seizures).
* Patient who will require fraction of inspired oxygen more than 0.6.
* Air leak from the chest tube.
* Patient with body temperature > 39 Celsius.
* Acute hepatitis or severe liver disease (Child-Pugh class C).
* Left ventricular ejection fraction less than 30%.
* Heart rate less than 50 beats/min.
* Second or third degree heart block.
* Systolic pressure < 90 mmHg despite of infusion of 2 vasopressors.
* Patients with known endocrine dysfunction.
* Patient with hypothermia
* Patient on Positive end expiratory pressure more than 14 cmH2o

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Resting energy expenditure after drug administration | The first baseline measurement will be taken before drug administration. The second measurement will be taken 24 hours after drug infusion.
  Resting energy expenditure will be measured using indirect calorimetry via metabolic module on General Electric ventilator

SECONDARY OUTCOMES:
Heart rate | 24 hours
  number of heart beats per minute
arterial blood pressure | 24 hours
  arterial blood pressure measured in mmHg
Richmond agitation and sedation scale | 24 hours
  range from -5 (unarousable) to +4 (combative)
Plasma interleukin-1β level | 24 hours
  determined by ELISA using a quantitative sandwich enzyme immunoassay technique
Tumor necrosis factor-α plasma concentration | 24 hours
  Enzyme immunoassay
partial pressure of oxygen in arterial blood | 24 hours
  the partial pressure of oxygen in arterial blood measured in mmHg
VO2 | 24 hours
  the oxygen consumption measured in mL/Kg/min
VCO2 | 24 hours
  carbon dioxide production measured in mL/Kg/min
end-tidal co2 | 24 hours
  the pressure of carbon dioxide in expired air measured in mmHg
cardiac output | 24 hours
  the amount of blood pumped by the heart during one minute

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdulatif, Professor, Study Chair — Professor and member of research committee of anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Walker RN, Heuberger RA. Predictive equations for energy needs for the critically ill. Respir Care. 2009 Apr;54(4):509-21. PMID 19327188
- [Background] Rubinson L, Diette GB, Song X, Brower RG, Krishnan JA. Low caloric intake is associated with nosocomial bloodstream infections in patients in the medical intensive care unit. Crit Care Med. 2004 Feb;32(2):350-7. doi: 10.1097/01.CCM.0000089641.06306.68. PMID 14758147
- [Background] Covelli HD, Black JW, Olsen MS, Beekman JF. Respiratory failure precipitated by high carbohydrate loads. Ann Intern Med. 1981 Nov;95(5):579-81. doi: 10.7326/0003-4819-95-5-579. PMID 6794409
- [Background] Fung EB. Estimating energy expenditure in critically ill adults and children. AACN Clin Issues. 2000 Nov;11(4):480-97. doi: 10.1097/00044067-200011000-00002. PMID 11288413